CLINICAL TRIAL: NCT02141360
Title: Advanced MRI Applications for Mild Traumatic Brain Injury - UCSF
Acronym: TBI-2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponser terminated early to start a larger feasability study
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 114-2014-GES-0001
Record Dates: First submitted 2014-05-12; First posted 2014-05-19 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Traumatic Brain Injury
Keywords: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Diagnostic mTBI (Experimental): MRI Diagnostic of subjects with mild Tramatic Brain Injury (mTBI)
  Interventions: Device: MRI Diagnostic
- Experimental: Diagnostic Non mTBI (Placebo Comparator): MRI Diagnostic of Non injured subjects that are closely matched to mTBI
  Interventions: Device: MRI Diagnostic

INTERVENTIONS:
Device: MRI Diagnostic — Commercially available MRI scanner using investigational or standard of care MR coils and a series of investigational Application Packs containing a predetermined set of MRI pulse sequences
  Other Names: Magnetic Resonance Image

SUMMARY:
This hypothesis-generating feasibility study compares mTBI Patients and Controls using advanced MRI Applications.

DETAILED DESCRIPTION:
This hypothesis-generating feasibility study is being conducted to determine potential associations between a broad range of clinical neurological symptoms and MR images, data, and clinical findings involved in mild traumatic brain injury (mTBI). These associations will be examined over the acute and sub-acute period (approximately 3 months) following injury to provide information useful for optimization of MR pulse sequences for mTBI applications.

The intent of this study is to broadly generate a range of potential mTBI biomarkers detectable using investigational MR pulse sequence technologies. Feasibility data attained in this study may be used for engineering program decision-making and in support of future scientific assessment, engineering development, published research databases or registries mTBI data and images, and other purposes determined by the Sponsor. The results of this study are not intended for use in regulatory submissions.

Subjects will be examined on commercially available MR scanners using investigational or standard of care MR coils and a series of investigational Application Packs containing a predetermined set of MR pulse sequences optimized by GEHC.

ELIGIBILITY:
Segment 1: Exclusion Criteria for mTBI subjects

Subjects will be excluded that have:

1. Loss of consciousness (LOC) ≥15 minutes;
2. Posttraumatic amnesia lasting ≥24 hr following a recent TBI event;
3. Diagnosis of moderate to severe TBI or GCS <13;
4. Structural brain injury indicated by previous neuroimaging findings;
5. Previous history of moderate to severe TBI;
6. Any previous history of mild TBI within the past 12 months;
7. Previously diagnosed brain white matter disease;
8. History of seizures within the past 10 years;
9. History of self-reported illicit drug abuse (except marijuana) in past 10 years;
10. History of alcohol abuse or dependence (per DSM-IV-TR Diagnostic Criteria);
11. Current primary Axis I or II psychiatric disorders, except for disorders classified as minor and not expected to impact study conduct or integrity (as detailed in Appendix F - Screening for Exclusion based on Axis I or II Disorders):
12. History of brain mass;
13. History of neurosurgery;
14. History of stroke;
15. History of dementia;
16. Known cognitive dysfunction;
17. Known structural brain disease or malformation;
18. Current anti-psychotic or antiepileptic medication usage;
19. That are unable or unwilling to complete study procedures accurately or have any conflict of interest that could affect study results, in the opinion of the investigator;
20. Contraindications to MRI scanning, including:

    1. Current or suspected pregnancy per site clinical practice;
    2. Other conditions that may constitute a hazard to the subject during study participation, determined by the investigator;
    3. Inability to comply with any part of the site's MR safety policy. 6.6. Segment 2 (non-TBI subject) Inclusion and Exclusion Criteria

Inclusion Criteria for Non-TBI subjects (Segment 2)

All included subjects will:

1. Aged ≥15 and ≤50 years old at the time of enrollment;
2. Be well matched to one or more mTBI patients in Segment 1, in the opinion of the Principal Investigator, with regards to:

   1. Age,
   2. Gender,
   3. Sociodemographic characteristics, and
   4. Handedness.
3. Be capable of sufficiently clear communication to allow the subject to provide written informed consent, or assent with parental or guardian consent for minors as described in Section 6.3 - Protection of Vulnerable Subjects, for participation in all parts of the study..

6.6.2. Exclusion Criteria for Non-TBI subjects (Segment 2)

Subjects will be excluded that:

1. Are currently pregnant based on subject self-report of pregnancy status;
2. Are currently enrolled in another Segment of this study;
3. Require medical care that would be adversely affected or delayed by participating, in the opinion of a physician investigator;
4. Prior diagnosis of mild TBI within the past 12 months;
5. Have structural brain injury indicated by previous neuroimaging findings;
6. Previous history of moderate to severe TBI within the past 10 years;
7. Previously diagnosed brain white matter disease;
8. History of seizures within the past 10 years;
9. History of illicit drug abuse (except marijuana) within the past 10 years
10. History of alcohol abuse or dependence (per DSM-IV-TR Diagnostic Criteria);
11. Current primary Axis I or II psychiatric disorders, except for disorders classified as minor and not expected to impact study conduct or integrity (as detailed in Appendix F - Screening for Exclusion based on Axis I or II Disorders):
12. History of brain mass;
13. History of neurosurgery;
14. History of stroke;
15. History of dementia;
16. Known cognitive dysfunction;
17. Known structural brain disease or malformation;
18. Current anti-psychotic or antiepileptic medication usage;
19. Have contraindications to MRI scanning, including:

    1. Current or suspected pregnancy per site clinical practice;
    2. Other conditions that may constitute a hazard to the subject during study participation, determined by the investigator;
    3. Inability to comply with any part of the site's MR safety policy.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Mukherjee, MD. PhD, Principal Investigator — University of California at San Francisco
Locations (1):
- University of California at San Francisco (UCSF), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Volunteer Control participants were scanned only for the purpose of operator training and calibrating the MRI device. No data was collected from these participants for the the purpose of analysis.
Groups:
- Experimental: Diagnostic mTBI: MRI Diagnostic of subjects with mild Traumatic Brain Injury (mTBI)
  MRI Diagnostic: Commercially available MRI scanner using investigational or standard of care MR coils and a series of investigational Application Packs containing a predetermined set of MRI pulse sequences
- Volunteer Controls: Non injured volunteers for device calibration
  Commercially available MRI scanner using investigational or standard of care MR coils and a series of investigational Application Packs containing a predetermined set of MRI pulse sequences
Period: Overall Study
Arm/Group | Experimental: Diagnostic mTBI | Experimental: Diagnostic Non mTBI | Volunteer Controls
Started | 11 | 6 | 6
Completed | 4 | 6 | 6
Not Completed | 7 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0
Not completed — Study Terminated before Visit | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Diagnostic mTBI | Experimental: Diagnostic Non mTBI | Total
Number analyzed (Participants) | 11 | 6 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 8 | 3 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: mTBI Progression Indicated by Clinical Neurological Characteristics, MRI Images, and Quantitative MRI Data From Novel Software
Description: To determine associations between clinical neurological data, MR images, quantitative data from novel software post-processing (sponsor developed software including Volumetry, Kurtosis, Resting State [RS], functional magnetic resonance imaging [fMRI], and additional post-processing modules may be provided
Time Frame: Baseline to 3 months
Population: Study was terminated and no subject outcome data were collected
Arm/Group | Experimental: Diagnostic mTBI | Experimental: Diagnostic Non mTBI | Volunteer Controls
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Experimental: Diagnostic mTBI | Experimental: Diagnostic Non mTBI | Volunteer Controls
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/11 | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Early termination of study due to limited recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No